CLINICAL TRIAL: NCT06941597
Title: Comparison of Two Gait Re-training Modalities During a Cardiac Rehabilitation Stay: Benefit of Orienteering Walking
Acronym: CAMCO
Status: Completed | Type: Observational
Sponsor: Fondation Ildys (Other)
Collaborators: Univ Brest, Laboratory ORPHY, F-29200 Brest, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RI2024_018
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases (CVD); Coronary Heart Disease (CHD); Heart Failure; Congenital Heart Disease
Keywords: cardiovascular diseases; cardiac rehabilitation; active walking; orienteering; heart rate
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac rehabilitation group: The management of patients included in this study is unchanged from that usually recommended. The patients included in the study will undergo the same rehabilitation sessions during their stay as patients coming to the centre as a matter of routine. In total, 3 sessions of active walking, 3 sessions of orienteering and 7 sessions of ergocycles were carried out during the stay. The cardiac rehabilitation programme lasted 3 weeks, and all the sessions evaluated as part of the study (active walking, orienteering and ergocycles) were carried out during the last two weeks of the rehabilitation course. For each activity (active walking and orienteering), a familiarisation session will be carried out before the session evaluated as part of the study. The order in which the orientation walking and active walking sessions are carried out will depend on the weeks in which the subjects are included, and may vary according to the organisation of the centre.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in France for women and the second leading cause of death for men after cancer. They cause around 140,000 deaths every year, or almost 400 people every day throughout France. CVD also accounts for over a million hospital admissions a year, 160,000 of which are attributable to heart failure.

At present, cardiovascular rehabilitation centres mainly use exercise training methods based on sessions on cycloergometers and active walking (walking on a track and/or treadmill). Convinced of the added value of Orienteering, we have included it in our routine treatment as part of our Cardiac Rehabilitation programme, in addition to sessions on cycloergometers and active walking since 2021. As there is little literature on the subject in our population of interest, the aim of this study is to provide evidence of the relevance of orienteering in the cardiac rehabilitation programme.

We hypothesise that orienteering induces a similar cardiac response, amount of physical activity and perception of symptoms compared with an active walking session, while providing greater enjoyment of the activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stabilised heart disease, coronary artery disease, heart failure, post-operative stay after cardiac surgery, congenital heart disease, patients at high cardiovascular risk and obliterative arteritis of the lower limbs;
* Who have been informed and do not object to the study;
* Over 18 years of age;
* Participating in a cardiac rehabilitation programme;
* With a walking distance of less than 3,600 metres;
* Able to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Persons under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are patients undergoing cardiac rehabilitation in the SSR cardiology department of the Ildys Foundation on the Ty Yann site.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-10-05 (Actual)

PRIMARY OUTCOMES:
To compare the average heart rate between an active walking session and an orientation walking session during the cardiac rehabilitation stay. | once during the second and third week of cardiac rehabilitation
  Average heart rate measured during the active walking session and the orienteering race.

SECONDARY OUTCOMES:
To compare the intensity of effort between the active walking, orienteering and cycloergometer sessions. | once during the second and third week of cardiac rehabilitation
  The maximum heart rate (bpm) will be collected for each of the three sessions.
To compare the intensity of effort between the active walking, orienteering and cycloergometer sessions. | once during the second and third week of cardiac rehabilitation
  The effort intensity score will be collected for each of the 3 sessions on a Borg scale (0-10). The modified Borg scale, also known as the CR10, is a simplified version of the original scale. It comprises 11 levels of perceived effort, ranging from 0 (no effort) to 10 (maximum effort).
Compare the performance of the physical activity performed during the active walking versus orienteering session. | once during the second and third week of cardiac rehabilitation
  Physical activity performance will be measured for each session by the total number of steps taken during active walking and orienteering.
Compare the performance of the physical activity performed during the active walking versus orienteering session. | once during the second and third week of cardiac rehabilitation
  Physical activity performance will be measured for each session by the time spent in the different intensity levels (light, moderate, vigorous) (in minutes and as a percentage).
Compare the performance of the physical activity performed during the active walking versus orienteering session. | once during the second and third week of cardiac rehabilitation
  Physical activity performance will be measured for each session by the distance covered in kilometres.
Compare the perception of effort between the active walking, orienteering and cycloergometer sessions. | once during the second and third week of cardiac rehabilitation
  Perceived motivation to carry out the activity using a Likert scale from 0 to 5. The Likert scale is a semantic scoring system, generally made up of 5 or 7 items, which is used in surveys to measure and evaluate perceptions, attitudes and opinions.
Compare the sensation of pleasure between the active walking, orienteering and cycloergometer sessions. | once during the second and third week of cardiac rehabilitation
  The feeling of pleasure for the three activity sessions will be measured on a Likert scale from 0 to 5. The Likert scale is a semantic rating system, generally composed of 5 or 7 items, which is used in surveys to measure and evaluate perceptions, attitudes and opinions.
To compare the desire to continue physical activity between the active walking, orienteering and cycloergometer sessions. | once during the second and third week of cardiac rehabilitation
  The desire to continue physical activity between the three physical activities will be measured by a Likert scale from 0 to 5. The Likert scale is a semantic rating system, generally composed of 5 or 7 items, which is used in surveys to measure and evaluate perceptions, attitudes and opinions.
Compare the heart rate kinetics during the three sessions (orienteering, active walking and cycloergometer). | once during the second and third week of cardiac rehabilitation
  Changes in heart rate over the three sessions (recorded every 5 minutes for 50 minutes for each session)

CONTACTS AND LOCATIONS:
Overall Officials: Klervie BAILLY, Principal Investigator — Fondation Ildys
Locations (1):
- Fondation ILDYS, Site de Ty Yann, Brest, France